CLINICAL TRIAL: NCT01668576
Title: Properties of Mesenchymal Stem Cells in Lung Transplant Candidates
Brief Title: Properties of Mesenchymal Stem Cells in Lung Transplant
Status: Terminated | Type: Observational
Why Stopped: Loss of funding
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, David C Neujahr, MD, Assistant Professor, Emory University
Other Study IDs: IRB00053075
Record Dates: First submitted 2012-08-15; First posted 2012-08-20 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Lung Transplantation
Keywords: mesenchymal stem cells; Lung transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — mesenchymal stem cells derived from subject bone marrow aspiration
Oversight: Data Monitoring Committee: No

SUMMARY:
The major limitation to long term survival in lung transplant recipients is the development of graft failure over time, termed bronchiolitis obliterans. The conventional therapies used to prevent rejection are not effective in preventing bronchiolitis obliterans. Therefore, new therapies are needed to address this problem. A growing body of research has focused on a unique population of bone marrow cells termed Mesenchymal Stem Cells (MSCs) to improve a range of medical conditions including heart failure, autoimmune disease, and inflammatory bowel disease. MSCs can prevent animal models of bronchiolitis obliterans. Because of this information, it is plausible that MSCs could help patients as a potential treatment in lung transplantation.

This proposal will test the immunologic properties of MSCs generated from such individuals to answer the question of whether generation of whether it would be feasible to use such cells in the future to prevent entities such as bronchiolitis obliterans.

The Investigator will approach patients who are being considered for a lung transplant because of end stage lung disease. Enrolled patients will undergo a bone marrow aspiration where a small amount of fluid is removed from their pelvic bone. Cells obtained in this procedure will be expanded in the Emory/Georgia Tech Cell Lab. MSCs will be expanded in this lab using cell culture conditions which are standardly used for MSCs.

DETAILED DESCRIPTION:
Problem of Interest: Lung transplantation represents a potential therapy for patients with end-stage lung diseases such as pulmonary fibrosis, emphysema and cystic fibrosis. The major limitation to long term survival in lung transplant recipients is the development of graft failure over time, termed bronchiolitis obliterans. The conventional therapies used to prevent rejection are not effective in preventing bronchiolitis obliterans. Therefore, new therapies are needed to address this problem. A growing body of research has focused on a unique population of bone marrow cells termed Mesenchymal Stem Cells (MSCs) to improve a range of medical conditions including heart failure, autoimmune disease, and inflammatory bowel disease. MSCs can prevent animal models of bronchiolitis obliterans. Because of this information, it is plausible that MSCs could help patients as a potential treatment in lung transplantation. MSCs can be obtained from 2 sources: commercially available MSCs which are generated from other normal volunteers and from the patient themselves. When MSCs are obtained from the patient for whom they are used, they are termed "autologous MSCs". A major potential drawback to the use of commercially available MSCs is that these cells contain proteins from other individuals which could provoke rejection when used in lung transplant recipients. Therefore, the use of autologous MSCs currently appears the most attractive option. What is not understood at the present time is the extent to which autologous MSCs obtained from chronically ill patients with end-stage lung disease still maintain properties which would be beneficial. This proposal will test the immunologic properties of MSCs generated from such individuals to answer the question of whether generation of whether it would be feasible to use such cells in the future to prevent entities such as bronchiolitis obliterans.

Overview on how this will be studied: The Investigator will approach patients who are being considered for a lung transplant because of end stage lung disease. Enrolled patients will undergo a bone marrow aspiration where a small amount of fluid is removed from their pelvic bone. Cells obtained in this procedure will be expanded in the Emory/Georgia Tech Cell Lab. MSCs will be expanded in this lab using cell culture conditions which are standardly used for MSCs. The Investigator will test the efficiency of expansion of these MSCs to determine if they can be obtained from all patients, or if there some patients demonstrate inefficient MSC expansion based on age or disease or other factors. The Investigator will then test in-vitro the ability of MSCs from different patients to prevent activation of the immune system when faced with proteins from other individuals. The Investigator believes this model system approximates the type of interaction that would occur if these MSCs were given to patients who received a lung transplant.

Benefit of research to knowledge and human health: It is not presently known whether patients with severe medical illness are able to have MSCs expanded. If it is found that MSCs can be readily obtained from such individuals and additionally find that such MSCs have properties which would be predicted to be beneficial in lung transplant, this study would provide the rationale to use MSCs as a therapeutic agent in patients undergoing lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 without regard to race or gender
* End stage lung disease from IPF, cystic fibrosis, emphysema, sarcoidosis or pulmonary hypertension
* Expected time from enrollment to transplant greater than 4 weeks
* Patient willing to undergo a bone marrow aspiration prior to transplantation

Exclusion Criteria:

* Patients under age 18
* Patients on significant immunosuppressive agents prior to transplant (specifically calcineurin inhibitors, cell cycle inhibitors or prednisone >0.5 mg/kg lean body weight)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant candidates
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Intrinsic variability of MSCs measured by time to third passage of confluent MSC | Post Co-Culture (24 hours)
  Assess for intrinsic variability of MSCs derived from individuals with end-stage lung disease across a range of ages, disease types, and comorbid conditions
2-3 IDO production measured as ug/mL of passage 3 MSCs | Post Co-Culture (24 hours)
  Demonstrate autologous MSCs have in-vitro immunoregulatory properties against allo-specific T cell responses and compare the MSC effects to conditioned media from MSCs
Percent specific inhibition of CD4 and CD8 T cell proliferation toward donor target cells in one way mixed-lymphocyte reactions | Post Co-Culture (24 hours)
  Test the immunoregulatory properties of MSCs in the setting of conventional levels of immune suppression

CONTACTS AND LOCATIONS:
Overall Officials: David Neujahr, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States